CLINICAL TRIAL: NCT02521090
Title: Targeting Recurrent Glioblastoma With Anti-CD3 x Anti-EGFR Bispecific Antibody Armed T Cells: A Phase I/II Study
Brief Title: EGFRBi-Armed Autologous T Cells in Treating Patients With Recurrent or Refractory Glioblastoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to lack of funding and a primary co-investigator of the trial leaving the institution.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sandeep Mittal, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-112; NCI-2015-00232 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-112 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Adult Brain Glioblastoma; Adult Gliosarcoma; Recurrent Brain Neoplasm
MeSH Terms: conditions — Gliosarcoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (EGFRBi-armed autologous T cells) (Experimental): PHASE I: Patients receive EGFRBi-armed autologous T cells IT twice weekly for 4 weeks.
  PHASE II: Patients receive EGFRBi-armed autologous T cells* IT twice weekly for 4 weeks and then IV over 15-30 minutes twice weekly for 2 weeks.
  *NOTE: Six selected patients receive EGFRBi-armed autologous T cells IV on day -3, -2, or -1 prior to first IT infusion.
  Interventions: Biological: EGFRBi-Armed Autologous T Cells; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: EGFRBi-Armed Autologous T Cells — Given IT and IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of epidermal growth factor receptor bispecific antibody (EGFRBi)-armed autologous T cells and how well it works in treating patients with glioblastoma that have come back or does not respond to treatment. EGFRBi-armed autologous T cells coated with antibodies (proteins used by the immune system to target and kill foreign objects such as cancer cells) may have great ability to seek out, attach to, and destroy glioblastoma cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) for 8 intrathecal (IT) injections (via lumbar puncture) of anti-cluster of differentiation (CD)3 × anti-EGFRBi armed activated T cells (aATC) (EGFRBi-armed autologous T cells) given twice per week for 4 weeks in a standard 3+3 dose escalation schema with 0.10, 0.50 and 1.00 × 10^9 EGFRBi-aATC per IT injection for a total of 0.8, 4.0, and 8.0 × 10^9 cells, respectively. (Phase I) II. To explore efficacy and confirm the toxicity profile of EGFRBi-aATC. (Phase II)

SECONDARY OBJECTIVES:

I. Measure immune responses in participants of the phase I/II trial by sequential monitoring of phenotype, interferon gamma (IFN-g) enzyme-linked immunoSpots (EliSpots), anti-glioblastoma (GBM) cytotoxicity of peripheral blood mononuclear cell (PBMC) (direct cytotoxicity against GBM cells) directed at GBM cell lines, T-helper 1 (Th1)/T-helper 2 (Th2) serum cytokine patterns, and anti-glioma antibodies in the cerebrospinal fluid (CSF)/serum during the "vaccinate and consolidate" process.

II. Assess survival and persistence of aATC in the CSF, and trafficking of IT-injected aATC out of the CSF into the bloodstream.

III. Image patients' brain with magnetic resonance imaging (MRI) (performed clinically in 2-month intervals; includes standard structural sequences and perfusion imaging) and alpha-[11C]methyl-L-tryptophan (AMT) positron emission tomography (PET) scan (under Wayne State University [WSU] Internal Review Board [IRB]/Karmanos Cancer Institute [KCI]-approved research protocol) before and after the aATC treatment regimen.

OUTLINE: This is a phase I dose-escalation study followed by a phase II study.

PHASE I: Patients receive EGFRBi-armed autologous T cells IT twice weekly for 4 weeks.

PHASE II: Patients receive EGFRBi-armed autologous T cells* IT twice weekly for 4 weeks and then intravenously (IV) over 15-30 minutes twice weekly for 2 weeks.

*NOTE: Six selected patients receive EGFRBi-armed autologous T cells IV on day -3, -2, or -1 prior to first IT infusion.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed intracranial glioblastoma or gliosarcoma (World Health Organization [WHO] grade IV) with evidence of clinical and radiographic (computed tomography [CT] or MRI brain) tumor progression (need not be biopsy proven)
* Patients who have undergone prior resection, radiation therapy, and/or chemotherapy (except bevacizumab)
* Karnofsky performance score >= 70 or Eastern Cooperative Oncology Group (ECOG) performance status = 0 or 1
* Patient agrees to undergo a baseline and a follow-up 11C-alpha-methyl-L-tryptophan (AMT)-PET scan during immunotherapy (IMT)
* No serious medical or psychiatric illness which prevents informed consent or intensive treatment is allowed
* Non pregnant: negative serum test for pregnancy, unless male, prior hysterectomy, tubal ligation, or postmenopausal; (Note: postmenopausal is defined as age > 55 with amenorrhea for > 1 year or age < 55 years with amenorrhea for 2 years and follicle stimulating hormone (FSH) level within postmenopausal range of institutional parameters; patients requiring FSH level to determine menopausal status need not have this performed and may choose to proceed with serum pregnancy testing)
* Required initial laboratory data (normal limits per treating institution; minor changes from the indicated laboratory guidelines will be allowed at the discretion of the treating team under special circumstances and reasons for the changes will be documented):
* Granulocytes >= 1,000/mm^3
* Absolute lymphocyte count >= 500/mm^3
* Platelet count >= 50,000/ul
* Hemoglobin >= 8 gm/dl
* Blood urea nitrogen (BUN) =< 1.5 times normal
* Serum creatinine < 1.8 mg/dl
* Creatinine clearance >= 50 ml/mm (can be calculated utilizing the Cockcroft & Gault equation)
* Bilirubin < 1.5 times upper limit of normal
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 times upper limit of normal
* Alkaline phosphatase < 5 times upper limit of normal
* Prothrombin time (PT) or international normalized ratio (INR) and activated partial thromboplastin time (aPTT) < 1.2 times upper limit of normal
* Negative human immunodeficiency virus (HIV)-1/2 serology
* Negative hepatitis B surface antigen
* Negative hepatitis C serology
* Left ventricular ejection fraction (LVEF) >= 45% at rest (multi gated acquisition [MUGA] or echocardiogram [ECHO])
* Each patient must be aware of the nature of their disease and must willingly consent to treatment after being informed of alternatives, potential benefits, side effects, and risks
* Surgery is done prior to IMT if needed for palliation, tumor debulking, pathological documentation of tumor recurrence; the patients may continue on study therapy even if they do not have measurable disease
* No other investigational agents, immunomodulating agents, or cancer chemotherapy are permitted for the duration and 12 months following the study IMT unless there is disease progression; radiotherapy is not permitted; appropriate antibiotics, blood products, antiemetics, fluids, electrolytes and general supportive care are to be used as necessary

Exclusion Criteria:

* Resective surgery within 2 months prior to the initial pre-treatment AMT-PET scan
* Severe increased intracranial pressure, status epilepticus, or other serious complications from the brain tumor, requiring emergency or urgent intervention
* Patients with a history of another malignancy within 5 years of study enrollment
* Patients with extracranial metastases
* Evidence of active bleeding or bleeding diathesis
* Patients will be ineligible for treatment on this protocol if (prior to protocol entry):

  * There is a history of a recent (within one year) myocardial infarction
  * There is a current or prior history of angina/coronary symptoms requiring medications and/or evidence of depressed left ventricular function (LVEF < 45% by MUGA or ECHO)
  * There is clinical evidence of congestive heart failure requiring medical management (irrespective of MUGA or ECHO results)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (Phase I) | Up to 7 days after the last infusion
Overall survival (OS) (Phase II) | From study enrollment to death due to any cause, assessed up to 2 years
  The median OS will be estimated with 95% confidence interval. Kaplan-Meier estimate of OS will be plotted. For quantitative measurements in immune evaluations, will calculate their means, standard deviations, medians, and examine the distributions of these data to ascertain whether normal theory methods are appropriate. Paired t-test or Wilcoxon signed-ranks test will be used for comparative analyses between each post-IMT time point versus pre-IMT.

SECONDARY OUTCOMES:
Change in cytokines profiles | Baseline to up to 1 year
  Mean, standard deviation, median and examine the distributions of these data will be calculated to ascertain whether normal theory methods are appropriate. Paired t-test or Wilcoxon signed-ranks test will be used for comparative analyses between each post-IMT time point versus pre-IMT. Bonferroni's adjusted p-values will be reported to control type I error rate. In addition, will assess the pattern of changes in the immune responses over time using graphical techniques such as LOWESS curves.
Changes in activated T cells | Baseline to up to 1 year
  Mean, standard deviation, median and examine the distributions of these data will be calculated to ascertain whether normal theory methods are appropriate. Paired t-test or Wilcoxon signed-ranks test will be used for comparative analyses between each post-IMT time point versus pre-IMT. Bonferroni's adjusted p-values will be reported to control type I error rate. In addition, will assess the pattern of changes in the immune responses over time using graphical techniques such as LOWESS curves.
Changes in cytotoxic T-lymphocyte as measured by IFN-gamma EliSpots directed at autologous tumor or GBM cell lines | Baseline to up to 1 year
  Mean, standard deviation, median and examine the distributions of these data will be calculated to ascertain whether normal theory methods are appropriate. Paired t-test or Wilcoxon signed-ranks test will be used for comparative analyses between each post-IMT time point versus pre-IMT. Bonferroni's adjusted p-values will be reported to control type I error rate. In addition, will assess the pattern of changes in the immune responses over time using graphical techniques such as LOWESS curves.
Changes induced by IMT | Baseline to up to 1 year
  Mean, standard deviation, median and examine the distributions of these data will be calculated to ascertain whether normal theory methods are appropriate. Paired t-test or Wilcoxon signed-ranks test will be used for comparative analyses between each post-IMT time point versus pre-IMT. Bonferroni's adjusted p-values will be reported to control type I error rate. In addition, will assess the pattern of changes in the immune responses over time using graphical techniques such as LOWESS curves.
Human anti-mouse antibody responses | Up to 1 year
  Serial serum samples will be tested and evaluated for the development of immunoglobulin G (IgG) and IgM anti-mouse antibody responses.
Peripheral blood measures | Up to 1 year

OTHER OUTCOMES:
Persistence of aATC in blood | Up to 1 year
  Will be evaluated whether the infused cells persist in vivo using fluorescence-activated cell sorting analysis for the mouse immunoglobulin G 2 alpha (IgG2a) (OKT3 part of the EGFRBi).

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Mittal, Principal Investigator — Barbara Ann Karmanos Cancer Institute